CLINICAL TRIAL: NCT04679220
Title: 36-Months Clinical Evaluation of Preheated Resin Composite
Brief Title: 36-Months Clinical Evaluation of Preheated and Room Temperature Resin Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 36.MCEPRCRCL
Record Dates: First submitted 2020-12-14; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Dental Leakage
Keywords: Resin Composite; Pain; Randomized Clinical Trial; Operative Dentistry; Preheating
MeSH Terms: conditions — Dental Leakage; Pain

STUDY DESIGN:
Intervention Model Description: One side of the mouth received preheated composite however in the other side the composite was placed in non-heated state following the manufacturer instructions.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-heated Resin Composite group (Active Comparator): Patients received Non-heated nanofilled resin composite on one side of the mouth
  Interventions: Procedure: Preheating
- Preheated Resin Composite group (Placebo Comparator): Patients received preheated nanofilled resin composite on the other side of the mouth
  Interventions: Procedure: Preheating

INTERVENTIONS:
Procedure: Preheating — For preheating RC prior to placement, a device called Therma-flo TM RC warming kit (Vista, Wisconsin, USA) was used according to manufacturer's instructions to preheat resin composites

SUMMARY:
Summary The aim of this study was to evaluate the effect of preheating resin composite (RC) on clinical performance of class I restorations in a period of 3-years using a split-mouth double-blinded randomized design.

DETAILED DESCRIPTION:
The description of the experimental design followed the Consolidated Standards of Reporting Trials (CONSORT) statement. The present study was a double-blinded (patients and examiner) randomized clinical trial anticipating the split mouth design. Thirty-five adult patients seeking dental treatment in Operative Department clinic at Faculty of Dentistry, University of Mansoura were enrolled in the current study with a total of 70 Class I restorations. No advertisement was made for participant recruitment, forming a sample of convenience. Each patient much sign a consent form before participating in the current study. The study was conducted from October 2017 to June 2020 as a part of Doctoral dissertation. Mansoura University institution's ethics committee approved the form and protocol before conducting the study. The sample size was calculated based on the clinical success rate (100% retention rate at 3 years) of posterior class I restorations restored with nanofilled composite observed in a previous study.28 According to several parameters including a significance level of 5%, the power of the test was calculated to be 80%, and equivalent limit of 15%. Upon these data, a sample size of 30 subjects was appropriate. Allowing for a 20% drop-out, sample size was set totalizing 35 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary caries involving occlusal surface only with ICDAS 2 and 3
* Patients with cavities no more than one-third of the intercuspal distance
* Patients must have a good oral hygiene;
* Patients with tooth gives positive response to testing with an electric pulp tester
* Patients with normal and full occlusion,
* Patients with opposing teeth should be natural with no restorations.

Exclusion Criteria:

* High caries risk patients with extremely poor oral hygiene,
* Patients involved in orthodontic treatment or periodontal surgery,
* Patients with periodontally involved teeth (chronic periodontitis)
* Patients with abutments should be excluded.
* Patients with heavy bruxism habits and clenching

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage % of patients with marginal staining | 3 years after restoration procedure
  Percentage of marginal staining in patients was clinically assessed using World Dental Federation FDI parameters using a scale from 1 to 5 scores (clinically very good, clinically good, clinically satisfactory, clinically unsatisfactory and clinically poor)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Statistical Analysis Plan can be shared to other researchers
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 3 Months for 3 years
Access Criteria: for anyone